CLINICAL TRIAL: NCT04703946
Title: Ankyloglossia in Neonates. Incidence of Short Sublingual Frenulum in Newborns at the Hospital Nostra Senyora de Meritxell. Relationship With Auxological Data, Associated Malformations or Diseases and Hereditary Component of the Newborn.
Brief Title: Incidence of Short Sublingual Frenulum in Newborns at the Hospital Nostra Senyora de Meritxell.
Status: Completed | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Francisco Guinot-Jimeno, Jefe departamento de odontopedaitria, Universitat Internacional de Catalunya
Other Study IDs: UIC-ODP-ANDORRA
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Ankyloglossia
MeSH Terms: conditions — Ankyloglossia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observacional — Analyze the incidence of short sublingual frenulum in newborns of the Hospital Nostra Senyora de Meritxell of the Principat of Andorra.
  1. Association or not of the AG with auxological parameters (weight, height, cranial perimeter) at birth.
  2. Association or not of the AG with sex.
  3. Association or not of the AG with gestational age.
  4. Association or not of the AG with other minor and major malformations.

SUMMARY:
The aim of the study was to analyze the incidence of short sublingual frenulum in newborns of the Hospital Nostra Senyora de Meritxell of the Principat of Andorra.

DETAILED DESCRIPTION:
Thus, the objective of this study was to determine the incidence of AG in newborns of the Hospital Nostra Senyora de Meritxell of the Principat of Andorra, as well as the relationship with auxological data, associated malformations or diseases and hereditary component of the newborn.

A random sample of 2167 individuals is enough to estimate, with a confidence of 95% and an accuracy of +/- 1 percentage units, a population percentage that is projected to be around 6%. The percentage of replenishment required is projected to be 0%. With this sample, it will be sufficient to estimate the children who have ankyloglossia, the % of relatives who also have it (a population percentage that is projected to be around 25%). Confidential and anonymous collection of data from patients' medical records for a period of 2 years and 8 months, and write them down in a database to finally correlate them and see if there is any association with the parameters studied.

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria are patients born from July 2018 to February 2021 (both inclusive) and of both genders.

Exclusion Criteria:

* The exclusion criteria are all those who were born abroad and who after 24 hours go to the Hospital of Andorra, those urgently transferred to other foreign centers after birth, as well as those who present medical records with lack of information.

Ages: 1 Minute to 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A random sample of 2167 individuals is enough to estimate, with a confidence of 95% and an accuracy of +/- 1 percentage units, a population percentage that is projected to be around 6%. The percentage of replenishment required is projected to be 0%.
Sampling Method: Probability Sample
Enrollment: 2167 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Ankilloglosia | 2 weeks
  presence or absence of Ankilloglosia

SECONDARY OUTCOMES:
type of short frenulum | 2 weeks
  One of the anatomical classification of the lingual frenulum is that of Coryllos, which classifies the lingual frenulum depending on its proximity to the lingual apex, based on 4 types

OTHER OUTCOMES:
height | 2 weeks
  height
weight | 2 weeks
  weight
cranial perimeter | 2 weeks
  cranial perimeter
sex | 2 weeks
  sex
type of lactation | 2 weeks
  type of lactation
hereditary factor (if the parents presented/present or not AG) | 2 weeks
  hereditary factor (if the parents presented/present or not AG)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No